CLINICAL TRIAL: NCT01604837
Title: The Optimal Oblique and Axial Angle of Fluoroscope for Superior Hypogastric Plexus Block
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Woo Seog Sim, Professor, Samsung Medical Center
Other Study IDs: 2012-03-074
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Pelvic Pain; Pelvic Malignancy; Superior Hypogastric Plexus Block
Keywords: superior hypogastric plexus block; pelvic malignancy; chronic pelvic pain

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pelvic malignancy group: those with diagnosis of gynecologic or urologic malignancy
- Pelvic chronic disease group: those with chronic pelvic pain with constitutional cause e.g. endometriosis

SUMMARY:
The recommended entry angle for superior hypogastric plexus block is different among references, and there is a need for suggesting a more accurate entry angle for this procedure. The investigators are trying to evaluate the entry angle for superior hypogastric plexus block by measuring these angle on the computed tomography image and apply these angle to the real patients.

DETAILED DESCRIPTION:
Superior hypogastric plexus block is a kind of sympathetic plexus block which are used to control the pelvic pain caused by malignancy or other chronic condition. Classic posterior approach for this procedure is inserting the block needle at L4 -5 level and proceed the needle 45 degrees medially and 30 degrees caudally to reach the target of anterolateral space of L5 - S1 intervertebral space. Waldman et al. introduced a different angle of 30 degrees medial and caudal with the same approach, while Stevens et al. recommended 15 degrees medial and 20 degrees caudal. As such, the recommended angle for this procedure is different among references, and there is a need for suggesting a more accurate entry angle for this procedure. Therefore, we are trying to evaluate the entry angle for superior hypogastric plexus block by measuring these angle on the computed tomography image and apply these angle to the real patients.

ELIGIBILITY:
Inclusion Criteria:

* Those undergoing abdominopelvic CT scan with pelvic malignancy or chronic pelvic pain with constitutional disease

Exclusion Criteria:

* Poor CT image with non-measurable axial or oblique entry angle

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those undergoing abdominopelvic CT scan with pelvic malignancy or chronic pelvic pain with constitutional disease
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the oblique entry angle | 1 month after abdominopelvic CT scan performed
  the oblique entry angle of superior hypogastric plexus block at L5-S1 level

SECONDARY OUTCOMES:
the axial entry angle | 1 month after abdominopelvic CT scan performed
  the axial entry angle of superior hypogastric plexus block at L4-S1 level

CONTACTS AND LOCATIONS:
Overall Officials: Woo Seog Sim, MD, PhD, Principal Investigator — Samsung Medical Center; Won Ho Kim, MD, Principal Investigator — Samsung Medical Center; Hye Won Song, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea